CLINICAL TRIAL: NCT02754973
Title: Effectiveness of an Integrated Experiential Training Program With Coaching by Nursing Students in Promoting Regular Physical Activity and Reducing Fatigue Among Childhood Cancer Patients
Brief Title: Integrated Experiential Training Program With Coaching by Nursing Students in Childhood Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW15-219
Record Dates: First submitted 2016-04-19; First posted 2016-04-28 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Child; Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): During hospitalization for cancer treatment, besides receiving usual care, participants in the experimental group will first receive a health education talk Participants will then be taught and encouraged to practice with some stretching and relaxing exercises during their hospitalization. After hospitalization, participants will receive an integrated experiential training program with coaching by nursing students through home visits.
  Interventions: Behavioral: an integrated experiential training program with coaching
- Placebo Control group (Placebo Comparator): Since participants in both groups are hospitalized in the same unit, to avoid contamination, participants in the placebo control group will receive the same intervention as those participants in the experimental group during their hospitalization. When discharged home, participants will receive an amount of time and attention (home visits by research assistants) that mimicked that received by the experimental group, but which is thought not to have any specific effect on the outcome measures.
  Interventions: Behavioral: Placebo Control

INTERVENTIONS:
Behavioral: an integrated experiential training program with coaching — The intervention will be implemented to each participant by a designated coach who is a trained nursing student during 28 home visits throughout a 6-month period (24 weeks) and each visit will last for about 1 hour. The 1-hour program consists of a 30-minute English tutorial session, and a 30-minute physical activity session with the coach. The same coach will pay a visit to a participant at twice a week for the first 4 weeks and then once a week for the subsequent 20 weeks. 4 levels of physical activity will be taught to the participants gradually according to their ability.
  Arms: Experimental group
Behavioral: Placebo Control — When discharged home, participants will receive an amount of time and attention (home visits by research assistants) that mimicked that received by the experimental group, but which is thought not to have any specific effect on the outcome measures. The placebo activities during the home visits may include playing cards or chess games, health advice on the prevention of influenza and healthy diet which will be conducted for 30 minutes.The participants will also receive a 30-minute English tutorial session with the research assistants in each home visit.
  Arms: Placebo Control group

SUMMARY:
Background: Despite the evidence that regular physical activity can have beneficial effects on the physical and psychological well-being of cancer patients, a review of the literature reveals that a majority of young cancer patients fail to attain the same levels of physical activity that they had before contracting the disease. There is scientific evidence that physical inactivity induces muscle catabolism and atrophy and cardiovascular diseases, which may lead to a further increase in fatigue and a decrease in the functional capacity of cancer patients. Empirical evidence is needed to explore an appropriate strategy for promoting physical activity in such patients.

Purposes: To examine the effectiveness of an integrated experiential training program with coaching by nursing students in promoting regular physical activity, reducing fatigue and enhancing quality of life among Hong Kong Chinese childhood cancer patients.

Design and Subjects: A randomised controlled trial (RCT), two-group pre-test and repeated post-test, within and between subjects design will be conducted. Recruitment of subjects will be carried out in a paediatric oncology ward of a Hong Kong acute care hospital.

Intervention: Participants in the experimental group will join an integrated experiential training program with coaching by nursing students, which contains 28 home visits by a designated nursing student as a coach for a 6-month period. Those in the placebo control group will receive an amount of time and attention (home visits by research assistants) that mimics that received by the experimental group.

DETAILED DESCRIPTION:
The aim of this study is to examine the effectiveness of an integrated experiential training program with coaching by nursing students in promoting regular physical activity, reducing fatigue and enhancing quality of life among Hong Kong Chinese childhood cancer patients.

Intervention

Experimental group

During hospitalization for cancer treatment, besides receiving usual care, a registered nurse will deliver participants a health education talk. Participants will then be taught and encouraged to practice some simple stretching and relaxing exercises. After discharged from the hospital, participants in the experimental group are scheduled to take part in an integrated experiential training program with coaching by nursing students. Each participant is allocated to a nursing student who was voluntarily trained as coaches for the program. The intervention is implemented to each participant by the designated coach during 28 home visits throughout a 6-month period (24 weeks) and each visit lasts for about 1 hour. The 1-hour program consists of a 30-minute English tutorial session, and a 30-minute physical activity session with the coach. The same coach pays a visit to a participant at twice a week for the first 4 weeks and then once a week for the subsequent 20 weeks. During the individual coaching sessions with the young people, the coaches will teach and demonstrate physical activities in 4 levels to the participants according to participants' ability.

Placebo control group

Since participants in both groups are hospitalized in the same unit, to avoid contamination, participants in the placebo control group will receive the same intervention as those participants in the experimental group during their hospitalization. When discharged home, participants will receive an amount of time and attention (home visits by research assistants) that mimicked that received by the experimental group, but which is thought not to have any specific effect on the outcome measures. The activities during the home visits over a six-month period include playing cards or chess games, health advice on the prevention of influenza and healthy diet which will be conducted for 30 minutes.The participants will also receive a 30-minute English tutorial session with the research assistants in each home visit.

To ensure the dosage of intervention delivered in terms of the amount, frequency, duration, and breadth would be adequate to assess physical activity levels, physical activity self-efficacy, cancer-related fatigue, depression, muscle strength, and quality of life, a research committee is crucial to assess the dosage of the intervention and to train the volunteer nursing students as coaches for the intervention. In particular, the safety and appropriateness of the intervention content were reviewed carefully by the committee before commencement. The members in the committee consist of an associate professor, an assistant professor and a research student from a local university who are equipped with extensive experience in conducting different research and particularly, psychosocial interventions for children with cancer. The committee also includes a professor in paediatric oncology and a specialist nurse with substantial experience in delivering care to children undergoing cancer treatment, and an assistant professor who is an expert specialising in sports and recreation management.

Data Collection Methods

Approval for the study was obtained from the hospital ethics committees. To identify potential subjects, the research student approach to eligible children and their parents after screening the medical records in a paediatric oncology ward of a public acute care hospital in Hong Kong. After explaining the study details, including its purpose, procedures and potential harms and benefits, parents allowing their children to take part are required to sign a consent form. In addition, the children who are going to participate are invited to write down their names on a specially designed child assent form and told that their participation is voluntary.

Data collection for the outcome variables is conducted at the time of the subject recruitment (T1), and six (T2), and nine (T3) months after the start of the intervention, except that physical activity levels of childhood cancer patients are collected at the time of the subject recruitment (T1), and nine (T2) months after the start of the intervention. Before randomisation, participants are required to complete the hand grip strength test with the hand-held dynamometers (HHD) and fill in a set of questionnaires including CUHK-PARCY, the Chinese versions of PA-SE, fatigue scale, CES-DC, and PedsQL cancer module. Semi-structured interviews will also be carried out.

Analysis

The Statistical Package for Social Sciences (SPSS) software, version 21.0 for Windows will be used to analyze quantitative data. Intention-to-treat analysis will be used and missing data will be substituted by the last-observation-carried-forward procedure. The comparability of the experimental and control groups will be assessed by using inferential statistics (independent t-test and chi-squared test). Descriptive statistics will be used to calculate the mean scores and standard deviation of different scales. Mixed between-within subjects ANOVA (split-plot ANOVA) and post-hoc analysis using the Tukey procedure will be used to determine whether the integrated experiential training program with coaching by nursing students was effective in reducing fatigue, increasing childhood cancer patients' levels of physical activity, self-efficacy and muscle strength, decreasing depressive symptoms and enhancing their quality of life. Descriptive phenomenology will be employed during the process of qualitative data analysis.

ELIGIBILITY:
Inclusion Criteria:

* aged between 9 to 18
* diagnosed with cancer at some time in the previous month and currently undergoing active treatments
* able to speak Cantonese and read Chinese

Exclusion Criteria:

* evidence of recurrence or second malignancies
* physical impairment or cognitive or learning problems identified from their medical records

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2015-05; Primary Completion 2017-08 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in levels of cancer-related fatigue from baseline at 9 month follow-up between intervention and control group | 9 month follow-up
  The primary outcomes are levels of cancer-related fatigue at 9 months after starting the intervention. The Chinese version of Fatigue Scale will be used to assess the fatigue of subjects.

SECONDARY OUTCOMES:
Levels of cancer-related fatigue at baseline | baseline
  The Chinese version of Fatigue Scale will be used to assess the fatigue of subjects.
Change in cancer-related fatigue from baseline at 6 month follow-up between intervention and control group | 6 month follow-up
  The Chinese version of Fatigue Scale will be used to assess the fatigue of subjects.
Levels of physical activity at baseline | baseline
  The Chinese University of Hong Kong: Physical Activity Rating for Children and Youth (CUHK-PARCY) will be used to assess the physical activity levels of the participants. It contains only one item which was derived from the Jackson Activity Coding and the Godin-Shephard Activity Questionnaire Modified for Adolescents. Participants will be asked to respond to the Chinese version of the CUHK-PARCY before randomization.
Levels of physical activity self-efficacy at baseline | baseline
  The Physical Activity Self-Efficacy (PA-SE) will be used to measure the children's self-confidence in their ability to participate in various age-appropriate physical activities. The PA-SE includes five items in which children are asked if they are 'not sure', 'a little sure' or 'very sure' that they can do such things as 'keep up a steady pace without stopping for 15-20 min'. Higher scores indicate higher self-efficacy. Participants will be asked to respond to the Chinese version of the PA-SE before randomization.
Change in levels of physical activity self-efficacy from baseline at 6 month follow-up | 6 month follow-up
  The Physical Activity Self-Efficacy (PA-SE) will be used to measure the children's self-confidence in their ability to participate in various age-appropriate physical activities. The PA-SE includes five items in which children are asked if they are 'not sure', 'a little sure' or 'very sure' that they can do such things as 'keep up a steady pace without stopping for 15-20 min'. Higher scores indicate higher self-efficacy. Participants will be asked to respond to the Chinese version of the PA-SE at 6 months after starting the intervention.
Change in levels of physical activity self-efficacy from baseline at 9 month follow-up | 9 month follow-up
  The Physical Activity Self-Efficacy (PA-SE) will be used to measure the children's self-confidence in their ability to participate in various age-appropriate physical activities. The PA-SE includes five items in which children are asked if they are 'not sure', 'a little sure' or 'very sure' that they can do such things as 'keep up a steady pace without stopping for 15-20 min'. Higher scores indicate higher self-efficacy. Participants will be asked to respond to the Chinese version of the PA-SE at 9 months after starting the intervention.
Depressive symptoms at baseline | baseline
  The depressive symptoms will be measured by the Centre for Epidemiological Studies Depression Scale for Children (CES-DC). It consists of 20 items in which cancer patients rated their experience of the previous 7 days on a 4-point Likert scale (0 = 'not at all', 1 = 'a little', 2 = 'sometimes', 3 = 'a lot'). The scores range from 0 to 60 with 16 as the cut-off score to represent a significant level of depression in the children. Higher scores corresponds to more number of depressive symptoms. Participants will be asked to respond to the Chinese version of the CES-DC before randomization.
Change in depressive symptoms from baseline at 6 month follow-up | 6 month follow-up
  The depressive symptoms will be measured by the Centre for Epidemiological Studies Depression Scale for Children (CES-DC). It consists of 20 items in which cancer patients rated their experience of the previous 7 days on a 4-point Likert scale (0 = 'not at all', 1 = 'a little', 2 = 'sometimes', 3 = 'a lot'). The scores range from 0 to 60 with 16 as the cut-off score to represent a significant level of depression in the children. Higher scores corresponds to more number of depressive symptoms. Participants will be asked to respond to the Chinese version of the CES-DC at 6 months after starting the intervention.
Change in depressive symptoms from baseline at 9 month follow-up | 9 month follow-up
  The depressive symptoms will be measured by the Centre for Epidemiological Studies Depression Scale for Children (CES-DC). It consists of 20 items in which cancer patients rated their experience of the previous 7 days on a 4-point Likert scale (0 = 'not at all', 1 = 'a little', 2 = 'sometimes', 3 = 'a lot'). The scores range from 0 to 60 with 16 as the cut-off score to represent a significant level of depression in the children. Higher scores corresponds to more number of depressive symptoms. Participants will be asked to respond to the Chinese version of the CES-DC at 9 months after starting the intervention.
Muscle strength at baseline | basline
  The right- and left-hand grip strengths of the participants were assessed by a dynamometer before randomization.
Change in muscle strength from baseline at 6 month follow-up between intervention and control group | 6 month follow-up
  The right- and left-hand grip strengths of the participants were assessed by a dynamometer 6 months after starting the intervention.
Change in muscle strength from baseline at 9 month follow-up between intervention and control group | 9 month follow-up
  The right- and left-hand grip strengths of the participants were assessed by a dynamometer 9 months after starting the intervention.
Levels of quality of life at baseline | baseline
  The Quality of life of the participants will be measured by the Chinese version of the PedsQL cancer module v. 3.0. This scale consists of 27 items which are categorized into eight different subscales, namely pain and hurt (2 items), nausea (5 items), procedural anxiety (3 items), treatment anxiety (3 items), worry (3 items), cognitive problems (5 items), perceived physical appearance (3 items) and communication (3 items). All items are evaluated on 5-point Likert scale by which the participants will be asked how much of a problem has been experienced over the last month. Participants will be asked to respond to the Chinese version of the PedsQL cancer module v. 3.0 before randomization.
Change in levels of quality of life from baseline at 6 month follow-up between intervention and control group | 6 month follow-up
  The Quality of life of the participants will be measured by the Chinese version of the PedsQL cancer module v. 3.0. This scale consists of 27 items which are categorized into eight different subscales, namely pain and hurt (2 items), nausea (5 items), procedural anxiety (3 items), treatment anxiety (3 items), worry (3 items), cognitive problems (5 items), perceived physical appearance (3 items) and communication (3 items). All items are evaluated on 5-point Likert scale by which the participants will be asked how much of a problem has been experienced over the last month. Participants will be asked to respond to the Chinese version of the PedsQL cancer module v. 3.0 at 6 months after starting the intervention.
Change in levels of quality of life from baseline at 9 month follow-up between intervention and control group | 9 month follow-up
  The Quality of life of the participants will be measured by the Chinese version of the PedsQL cancer module v. 3.0. This scale consists of 27 items which are categorized into eight different subscales, namely pain and hurt (2 items), nausea (5 items), procedural anxiety (3 items), treatment anxiety (3 items), worry (3 items), cognitive problems (5 items), perceived physical appearance (3 items) and communication (3 items). All items are evaluated on 5-point Likert scale by which the participants will be asked how much of a problem has been experienced over the last month. Participants will be asked to respond to the Chinese version of the PedsQL cancer module v. 3.0 at 9 months after starting the intervention.
Change in levels of physical activity from baseline at 9 month follow-up between intervention and control group | 9 month follow-up
  The Chinese University of Hong Kong: Physical Activity Rating for Children and Youth (CUHK-PARCY) will be used to assess the physical activity levels of the participants. It contains only one item which was derived from the Jackson Activity Coding and the Godin-Shephard Activity Questionnaire Modified for Adolescents. Participants will be asked to respond to the Chinese version of the CUHK-PARCY at 9 months after starting the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lam KKW, Li WHC, Chung OK, Ho KY, Chiu SY, Lam HS, Chan GCF. An integrated experiential training programme with coaching to promote physical activity, and reduce fatigue among children with cancer: A randomised controlled trial. Patient Educ Couns. 2018 Nov;101(11):1947-1956. doi: 10.1016/j.pec.2018.07.008. Epub 2018 Jul 7. PMID 30007765